CLINICAL TRIAL: NCT03726632
Title: Causality of Poisoning of the Elderly: Prospective Study Based on Data From the Poison Control Centre of Bordeaux Over 5 Months
Brief Title: Causality of Poisoning of the Elderly: Prospective Study Based on Data From the Poison Control Centre of Bordeaux
Acronym: GERIATOX
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2017/02
Record Dates: First submitted 2018-10-12; First posted 2018-10-31 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Intoxication
Keywords: Elderly; Intoxication; Poison Control centre; Poisoning; Accidental exposure; Prevention
MeSH Terms: conditions — Poisoning

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Elderly is often associated with social, physiological and psychic changes. However, no study has examined accidental poisoning-induced changes.

The objective of the study is to identify and analyze the various causes of potentially toxic accidental exposure of the elderly to determine preventable causes and propose prevention strategies.

DETAILED DESCRIPTION:
Elderly is often associated with social, physiological and psychic changes. Many studies tried to demonstrate their influence in the genesis of pathological events such as falls or suicide of the elderly but none on the genesis of accidental poisoning.

However, poisoning in this age group is frequent and sometimes severe. In order to improve care of the elderly, it seems necessary to focus on potential toxic accidental exposure.

For this, Poison Control Centre of the University Hospital of Bordeaux has identified the causes over a period of 5 months (from 01 March to 31 July 2017) from calls to the centre.

ELIGIBILITY:
Inclusion Criteria:

* All subjects aged 65 and over,
* Victims of accidental exposure regardless of the agent (drug, household product, plant ...)
* Victims of voluntary exposure (out of suicidal behavior)
* And for which a call (notice, report) to the Poison Control Centre of Bordeaux has been recorded.
* Calling dates between March 1st and July 31st, even if the exhibition is prior to March 1st, 2017).

Exclusion Criteria:

* Suicide
* Calls for inquiries

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All subjects aged 65 and over, victims of accidental or voluntary (excepted suicide) exposure of an agent (drug, household product, plant ...) and for who a call the Bordeaux Poison Control Centre has been called.
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2017-08-02 (Actual); Study Completion 2017-08-02 (Actual)

PRIMARY OUTCOMES:
Nature of the agent | Baseline
  The nature of the agent has to be chosen among (1 choice only): drug, chemical, household product, DIY product, phytosanitary product, gas, plant, foreign body, food

SECONDARY OUTCOMES:
Circumstance of the event | Baseline
  The circumstance of the event has to be chosen among (1 choice only): accidental / voluntary
Exposition route of exposure | Baseline
  The exposition route of exposure has to be chosen among (1 choice only): ingestion, eyepiece, dermal, inhalation or multiple routes
symptoms | Baseline
  Number / Nature
Poisoning Severity | Baseline
  The poisoning severity is evaluated using the Poisoning Severity Scale (PSS score). Severity grades: None (No symptoms or signs related to poisoning); MINOR (Mild, transient and spontaneously resolving symptoms); MODERATE (Pronounced or prolonged symptoms); SEVERE (Severe or life-threatening symptoms); DEATH
Death | Baseline
  death before the call
Frailty status | Baseline
  The frailty status is calculated from the following factors: sensory disturbance, cognitive and/or neurological disorder, psychiatric disorder, autonomy / dependence, concomittant treatments
packaging of the agent | Baseline
  The packaging of the agent has to be chosen among (1 choice only): solid, liquid, gaseous, powder and if drug: tablet, drops, syrup, patch, injectable
Concomittant treatment | Baseline
  Number of prescription drugs

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Anti Poision du CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No